CLINICAL TRIAL: NCT02943382
Title: The Use of Fingerprick Autologous Blood (FAB) in the Treatment of Mebomian Gland Dysfunction (MGD)
Brief Title: Fingerprick Autologous Blood (FAB) in Mebomian Gland Dysfunction (MGD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bedford Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 473/2016/301
Record Dates: First submitted 2016-08-12; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Disease
Keywords: MGD; Autologous Serum; Meibomian gland dysfunction; Dry eye disease; FAB; Fingerprick autologous blood
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

ARMS (1):
- Fingerprick Autologous Blood (FAB) (Experimental): Assigned treatment with FAB
  Interventions: Other: Fingerprick autologous blood (FAB)

INTERVENTIONS:
Other: Fingerprick autologous blood (FAB) — Pricking of cleaned finger using diabetic lancet and applying blood droplet to affected eye. Repeated with separate finger for other affected eye.

SUMMARY:
Dry eye disease remains one of the most common complaints seen in ophthalmic clinics. Causes of dry eye are multifactorial, with the most common cause of evaporative dry eye disease being meibomian gland dysfunction (MGD).

Fingerprick autologous blood (FAB) is a novel method which uses a patient's own blood to treat dry eye conditions.

DETAILED DESCRIPTION:
Dry eye disease remains one of the most common complaints seen in ophthalmic clinics, with one in four patients reporting symptoms of the condition (including soreness, foreign body sensation or temporary blurring of vision). Causes of dry eye are multifactorial, with the most common cause of evaporative dry eye disease being meibomian gland dysfunction (MGD).

A chronic, abnormality of the glands lining the eyelid. MGD results in alteration of the tear film, symptoms of eye irritation, inflammation and ocular surface disease. In those with moderate or severe disease (as defined by symptoms, clinical signs and corneal staining), anti-inflammatory therapy is recommended, with topical steroids or oral tetracyclines. However, both these treatments are accompanied by side effects; topical steroids cause increased intraocular pressure, and predispose to eye infection and cataracts, whilst tetracyclines cause skin phototoxicity.

Autologous serum drops are used as a treatment for severe dry eyes by providing growth factors and anti-inflammatory mediators to the ocular surface. It is derived from the liquid component of blood, after clotting factors and blood cells have been extracted. Obtaining this carries its own problems: numerous venesections from the patient, fridge storage to prevent bacterial contamination, and individual funding request as it is expensive.

The growth factors and anti-inflammatory mediators in serum are also present in whole blood; which can be obtained using a finger prick technique as in diabetics, thus bypassing the cost and storage problems associated with autologous serum.

Finger prick autologous blood (FAB) has shown efficacy and safety in the treatment of severe dry eye syndrome patients and persistent corneal epithelial defects. In this study, the investigators aim to find out whether FAB is an effective alternative to long-term anti-inflammatories in the treatment of MGD. Patient's with MGD will be recruited from Moorfields Eye clinic at Bedford Hospital. The study will be conducted over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with meibomian gland dysfunction (based upon lid margin signs and consequent dry eye syndrome) with discomfort which affects their daily life, and who want further treatment and remain symptomatic despite optimum treatment (lid hygiene and massage, tried or are on artificial lubricants at least four times a day and tried or are on oral omega-3 oils).

Exclusion Criteria:

* Patients who do not have capacity to consent • Children (under 18 years old)
* Infected finger or systemic infection or on systemic antibiotics for infection
* Patients with immunodeficiency
* Infected finger or systemic infection or on systemic antibiotics for infection.
* Patients with active microbial infection, acute herpes simplex or herpes zoster keratitis, drug toxicity, vitamin A deficiency, or recurrent corneal erosion.
* Past Ophthalmic history of corneal transplantation.
* Pregnant or breast feeding women
* Fear of needles and unwillingness to carry out repeated finger pricks
* Past or current ocular malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in clinical symptoms assessed using the OSDI questionnaire | 2 months
  Ocular surface disease index questionnaire (OSDI)

SECONDARY OUTCOMES:
Improvement of Meibomian Gland Dysfunction signs assessed using the International Workshop on Meibomian Gland Dysfunction report on grading criteria | 2 months
  To improve signs (grading of MGD) as per 'The International Workshop on Meibomian Gland Dysfunction' report on grading criteria (Tomlinson, 2011)

IPD SHARING:
Plan to Share IPD: Undecided